CLINICAL TRIAL: NCT00187889
Title: A Double-Blind, Multicenter, Placebo Controlled Study of Aldosterone Blockade (Eplerenone) in Women With Chest Pain, Coronary Vascular Dysfunction and Evidence of Myocardial Ischemia in the Absence of Significant Epicardial Coronary Artery Disease
Brief Title: EWISE: Study of Eplerenone in Women With Chest Pain, Coronary Vascular Dysfunction and Evidence of Myocardial Ischemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EWISE; R01 H267173-01
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Results first posted 2013-10-14 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2011-10

CONDITIONS: Ischemic Heart Disease
Keywords: Microvascular Disease; Women; Ischemic Heart Disease; WISE
MeSH Terms: conditions — Myocardial Ischemia | interventions — Eplerenone; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eplerenone (Active Comparator): Eplerenone 25 mg (1 pill)daily for 1 week then uptitrated to 50 mg (2 pills)daily for 15 weeks.
  Interventions: Drug: Eplerenone
- Placebo or sugar pill (Placebo Comparator): Placebo blinded as 25 mg tablet once daily for 1 week then uptitrated to 2 pills daily for 15 weeks.
  Interventions: Drug: Placebo or sugar pill

INTERVENTIONS:
Drug: Eplerenone — Eplerenone 25 mg (1 pill) daily for 1 week then uptitrated to 50 mg (2 pills) daily for 15 weeks.
  Arms: Eplerenone
Drug: Placebo or sugar pill — Placebo blinded as 25 mg tablet(1 pill) once daily for 1 week then uptitrated to 50 mg (2 pills) daily for 15 weeks.
  Other Names: Placebo
  Arms: Placebo or sugar pill

SUMMARY:
Some women have chest pain even without having a blockage in one of the major blood vessels that supplies blood to the heart. In many of these women the microscopic (small) blood vessels in the heart do not function normally. This study seeks to determine if treatment with eplerenone, a commercially available diuretic, can improve the function of these microscopic blood vessels and, possibly, improve the chest pain.

DETAILED DESCRIPTION:
INDICATION: Coronary Vascular Dysfunction (Endothelial Dysfunction and/or Microvascular angina).

OBJECTIVES: To investigate effects of aldosterone blockade (eplerenone) on coronary vascular function.

PATIENT POPULATION: Women who meet the National Heart, Lung and Blood Institute-sponsored WISE (Women Ischemia Syndrome Evaluation) study criteria of chest discomfort, coronary vascular dysfunction and undergoing evaluation for myocardial ischemia in the absence of significant coronary artery stenosis.

STUDY DESIGN: A prospective, randomized, double blind placebo-controlled, comparative trial of eplerenone, given in the presence of a renin-angiotensin blocker (ACE-I or ARB in the case of ACE-I intolerance).

TREATMENT: Eplerenone 25mg titrated to 50mg as tolerated per day versus placebo for four months

PRIMARY EFFICACY PARAMETER(S): Epicardial coronary artery endothelial function at Week 16 (adjusted for baseline treatment group and site by treatment interaction variables) comparing the eplerenone group to the placebo group.

SECONDARY EFFICACY PARAMETERS: Microvascular coronary endothelial function at Week 16 (adjusted for baseline treatment group and site by treatment interaction variables) comparing the eplerenone group to the placebo group.

OTHER EFFICACY PARAMETERS:

* Coronary flow reserve
* Chest discomfort as measured by the Seattle Angina Questionnaire
* DASI

SAFETY PARAMETERS: Blood pressure, pulse rate and frequency and occurrence of adverse events. The latter will include serum K and Creatinine.

STATISTICAL RATIONALE AND ANALYSIS: A statistical rationale for the number of patients in the study has been provided. Interim analyses are planned after 10 patients have completed treatment in each group.

ANTICIPATED TOTAL NUMBER OF PATIENTS: 50 (25 per treatment group).

ANTICIPATED NUMBER OF PATIENTS AT EACH SITE: Approximately 13.

PARTICIPATING SITES: University of Florida (Carl Pepine, MD), Emory University (Arshed Quyyumi, MD), Rhode Island Hospital (Barry Sharaf, MD), and Mayo Clinic (Amir Lerman, MD). There is an existing relationship between the first 3 sites and the Mayo Clinic site is familiar with all necessary protocol procedures and is anxious to participate. The University of Florida will serve as the main contracting site.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant women with chest discomfort who are 21 to 75 years of age and from diverse racial/ethnic groups.
* Suspected ischemic heart disease (IHD) but no severe coronary stenosis (> 50% diameter reduction) on coronary angiography used to qualify for WISE.
* Endothelial dysfunction, defined as failure to dilate to intracoronary acetylcholine (< 5% increase in mean lumen diameter).
* If possible, patients should be taking stable, maximally tolerated dose of either an angiotensin-converting enzyme inhibitor [ACEI] (or an angiotensin II receptor blocker [ARB] if ACEI intolerant)

Exclusion Criteria:

* Women who are breast-feeding or who are pregnant. Women of childbearing potential may be enrolled but must agree not to become pregnant during the course of the study and must practice a method of birth control considered reliable by the investigator. If established on hormonal contraceptives for more than 3 months, patients will be allowed to participate provided that this therapy remains constant throughout the study. If a patient becomes pregnant or begins breast-feeding during the study, she must be withdrawn immediately.
* Acute ischemic syndrome defined as acute myocardial infarction [MI] (by enzyme or electrocardiogram [ECG] criteria) or unstable angina within 1 month of entry.
* Uncontrolled moderate hypertension: sitting blood pressure > 160/95mmHg with measurements recorded on at least 2 occasions (for blood pressure control patients must first be stabilized, preferably with a diuretic, and remain on that dosing regimen throughout participation in the study).
* Severe heart failure defined as New York Heart Association (NYHA) Class III or IV on treatment.
* Coronary revascularization by either coronary artery bypass grafting (CABG) or percutaneous transluminal coronary angioplasty (PTCA) or stent placement.
* Conditions likely to influence outcomes independent of IHD: severe lung, renal (creatinine >1.8 or creatinine clearance [CrCl] ≤ 50ml/min) or hepatic disease; surgically uncorrected significant congenital or valvular heart disease; and other diseases likely to be fatal or require frequent hospitalizations within the next six months.
* Adherence or retention reasons: recent alcoholism or drug abuse; psychiatric illness including severe depression; dementia; active participation in any other research trial other than WISE; or unwilling to complete follow-up evaluations including repeat testing.
* Hypersensitivity to any medications to be used in the study
* Documented obstructive hypertrophic cardiomyopathy.
* Aortic stenosis (valve area < 1.5cm).
* Left ventricular (LV) dysfunction (ejection fraction <= 35%).
* History of significant cocaine or amphetamine abuse.
* Serum potassium > 5.0meq/l at baseline
* Taking potent CYP3A4 inhibitors (ketoconazole, itraconazole, nefazodone, troleandomycin, clarithromycin, ritonavir, nelfinavir)
* Intolerance to ACEI and ARB medications
* Use of potassium supplements or potassium sparing diuretics

Ages: 21 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2004-08; Primary Completion 2009-02 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl J Pepine, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Derived] Bavry AA, Handberg EM, Huo T, Lerman A, Quyyumi AA, Shufelt C, Sharaf B, Merz CN, Cooper-DeHoff RM, Sopko G, Pepine CJ. Aldosterone inhibition and coronary endothelial function in women without obstructive coronary artery disease: an ancillary study of the national heart, lung, and blood institute-sponsored women's ischemia syndrome evaluation. Am Heart J. 2014 Jun;167(6):826-32. doi: 10.1016/j.ahj.2014.01.017. Epub 2014 Mar 1. PMID 24890531

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants was recruited into the study by using flyers, and asked about interest in the medical clinics.
Pre-assignment Details: A total of 70 participants were screened for the study. Out of the 70 participants a total of 18 screened failed, 1 patient was withdrawn due to developing a spasm during the provocative testing screening which was believed to represent thrombosis and was not randomized to the study.
Period: Overall Study
Arm/Group | Eplerenone | Placebo or Sugar Pill
Started | 25 | 26
Completed | 19 | 22
Not Completed | 6 | 4
Not completed — Withdrawal by Subject | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Epleranone: Epleranone 25 mg daily for 1 week then uptitrated to 50 mg daily for 15 weeks.
- Total: Total of all reporting groups
Arm/Group | Epleranone | Placebo or Sugar Pill | Total
Number analyzed (Participants) | 25 | 26 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 22 | 44
  >=65 years | 3 | 4 | 7
Age Continuous [Mean (Standard Deviation); unit: years] | 53 (9) | 54 (11) | 53 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 51
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 26 | 51

OUTCOME MEASURES:

1. Primary Outcome: Epicardial Coronary Artery Endothelial Function (Adjusted) at Week 16 Comparing the Eplerenone Group to the Placebo Group
Description: The primary measure was the relative change in coronary diameter to acetylcholinem (ACH) at 16 weeks adjusted for baseline reactivity to acetylcholine. Change in coronary artery diameter after ACH was measured in mm at baseline and 16 weeks. Percent change at 16 weeks - percent change at baseline was the outcome.
Time Frame: 16 weeks
Population: power analysis: Study planned to detect a 12% difference in change from baseline to 16 weeks between treatment groups (SD=14%), in the primary outcome leading to a planned sample size of 22 per group (44 total) for 80% power, P=0.05 2-sided. Study allowed for 6 dropouts, leading to a final N=50 planned (25 per group). Per protocol analysis used.
Measure: Mean (Standard Deviation); unit: % change wk16-%change wk0- unitless
Groups:
- EPLERINONE: Active drug
- PLACEBO: Inert Placebo
Arm/Group | EPLERINONE | PLACEBO
Number analyzed (Participants) | 19 | 22
% change wk16-%change wk0- unitless | -1.2 (15.4) | -10.7 (25.6)
Statistical Analysis 1: Comparison: EPLERINONE vs PLACEBO; The null hypothesis is that the treatments are equivalent with respect to the primary outcome. The Satterthwaite corrected t-tests adjusts for potentially unequal variance in the groups; Test type: Superiority or Other; p = 0.15, Satterthwaite corrected t-test — The P-value applies to this comparison, without adjustment, to the completers of the trial; Mean Difference (Net) = -9.6, 95% CI 2-sided [-22.8 to 3.6], Standard Error of Mean 6.7 — An expanded definition of the outcome measure is the difference between the percentage change (week 16) and the percentage change week 0). This is a calculation based on 4 measurements
Statistical Analysis 2: Comparison: EPLERINONE vs PLACEBO; The null hypothesis is that treatments are equivalent on this outcome. The study was powered around the primary outcome. No adjustment for multiple comparisons was planned; Test type: Superiority or Other; p = 0.92, Satterthwaite corrected t-test; Mean Difference (Net) = -0.04, 95% CI 2-sided [-0.79 to 0.72], Standard Error of Mean 0.39 — The Satterthwaite corrected t-tests adjusts for potentially unequal variance in the groups. This is a different outcome variable than the primary

2. Secondary Outcome: Microvascular Coronary Flow Reserve(Adjusted) at Week 16 Adjusted for Baseline Coronary Flow Reserve Comparing the Eplerenone Group to the Placebo Group
Description: Coronary flow reserve is a ratio of coronary blood flow velocity before and after adenosine. The outcome measure is the difference between the coronary flow reserve at 16 weeks adjusted for coronary flow reserve at baseline.
Time Frame: 16 weeks
Population: See Primary Outcome. The studied was only powered for the primary outcome. All completers are included per protocol analysis.
Measure: Mean (Standard Deviation); unit: difference of ratios (unitless)
Groups:
- EPLERENONE: Active Drug
Arm/Group | EPLERENONE | PLACEBO
Number analyzed (Participants) | 13 | 18
difference of ratios (unitless) | -0.4 (0.9) | -0.4 (1.2)

ADVERSE EVENTS:
Arm/Group | Epleranone | Placebo or Sugar Pill
Serious Adverse Events (participants affected / at risk) | 1/24 | 0/26
Other Adverse Events (participants affected / at risk) | 3/24 | 3/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epleranone (N=24) | Placebo or Sugar Pill (N=26)
Deep venous thrombosis (Vascular disorders) | 1 (1) | 0 (0) — Day 17 hospitalized for DVT, anticoagulated with coumadin,recovered uneventfully. DVT occurred in the leg that cath was performed consider possible related, patient on placebo.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epleranone (N=24) | Placebo or Sugar Pill (N=26)
chest pain (Cardiac disorders) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No